CLINICAL TRIAL: NCT04284176
Title: Influence of the Quality of Movement in the "Non-use" of the Upper Extremity Affected in Children Hemiparesis: Mirror Therapy and Action-observation as Therapeutic Strategies
Brief Title: Movement in the Non-use of the Affected Upper Extremity in Children Hemiparesis: Mirror Therapy and Action-observation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEUSPU
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-02

CONDITIONS: Hemiplegia, Infantile
MeSH Terms: conditions — Hemiplegia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirrow therapy and action-observation therapy (Experimental): The intervention include 20 hours, applied during a four-week period (1 hour per day from Monday to Friday) at home. The first 15 minutes will include myrror therapy 6 activities and the remaing 45 minutes both unimanual and bimanual action-observation therapy activities.
  Interventions: Other: Mirror therapy and action-observation therapy
- Action-observation therapy (Experimental): The intervention include 20 hours, applied during a four-week period (1 hour per day from Monday to Friday) at home. There protocol includes both unimanual and bimanual action-observation therapy activities.
  Interventions: Other: Mirror therapy and action-observation therapy

INTERVENTIONS:
Other: Mirror therapy and action-observation therapy — The mirror therapy and action-observation therapy group will receive for 20 days a daily therapy of 15 minutes at home of MT and 45 of AOT, whereas the action-observation therapy group will receive 60 minutes of AOT.

SUMMARY:
Children with cerebral palsy hemiplegia present a restriction in the daily activities due to the limitation in the active movement of the affected upper extremity.

The mirror therapy (MT) in children with hemiparesis produces an improvement in the quality of movement and in the perception of the affected upper extremity. The action-observation therapy (AOT) favors the motor behaviour of the affected upper extremity through the observation of sequences of systematic activities and their posterior execution. It also produces an increase in the excitability of the corticospinal tract, originating muscular pattern contraction similar to the observed ones and favoring the motor activity.

The combination of both therapies might improve the quality of movement of the upper extremity and provide a major cortical activation and increase the spontaneous use on having created the only protocol of intervention which includes the benefits of both interventions.

The principal aim of this study is to analyze the influence of the quality of movement in the spontaneous use of the upper extremity affected in children with hemiparesis as well as the improvement of both variables across MTAO. Another specific aim will be to determine if "the non-use" is determined by the quality of the movement of the segment, if the MTAO reduces "the non-use" of this extremity as well as to obtain a protocol of intervention that increases the quality of movement and the spontaneous long-term use.

A randomized controlled trial will be carry out in children with hemiparesia between 6 and 12 years, with a spontaneous use of the hand according to the scale HOUSE, a level Manual Ability Classification System (MASC) I-III and a good cooperation and cognition. Those with a severe spasticity, previous surgery of the upper extremity and the use of botox will be excluded. The children will be divided in two groups. The experimental group will receive for 20 days a daily therapy of 15 minutes at home of MT and 45 of AOT, whereas the control group will receive 60 minutes of AOT.

Four measurements will be obtained: basal situation, at the end of the treatment and measures of follow-up to 3 and 6 months after the end of the treatment. Despite the sociodemographic variables, measures of the quality of the movement, the spontaneous use of the upper extremity, the questionnaire CHEQ and the AHA scale.

DETAILED DESCRIPTION:
Two protocols are designed to be carried out at home. The AOT protocol includes 15 set of daily life upper limb uni/bimanual activities (8 sets for bimanual activities and 7 sets for unimanual activities).

The MTAO group include 6 mirror therapy activities and the same activities that are included in the AOT protocol.

A pilot study will be conducted for sample size calculation, assessing the AHA and Jebsen-Taylor scales, before and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children with hemiparesia.
* From 6 to 12 years,
* A spontaneous use of the hand according to the scale HOUSE, a level MACS I-III
* A good cooperation and cognition

Exclusion Criteria:

* Severe spasticity
* Previous surgery of the upper extremity
* The use of botox

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the affected hand and arm in bimanual performance assess by Assisting Hand Assessment (AHA) scale | 6 months
  AHA scale includes several domains: general use, arm use, grasp-release, fine motor adjustments, coordination and rhythm. 22 items are scored and converted to 0-100 logit-based AHA units.
Functionality of the affected hand assess by Jensen-Taylor scale | 6 months
  The Jebsen-Taylor scale includes 7 subtests: writing, card turning, picking up small objects, stacking checkers, stimulated feeding, moving lights objects, moving heavy objects. Normative data are described for adults, but not for children.
Experience of children in the use of the affected hand during activities where two hands are usually required assess by the Children's Hand-use Experience Questionnaire (CHEQ). | 6 months
  The CHEQ questionnaire ask about some activities that typically require the use of both hands. The results are converted into logits using Rasch analysis.
Grip strength assess by hand grip dynamometer | 6 months
  Hand grip dynamometer
Muscular activity of the wrist muscles assess by Surface electromyography (EMG) | 6 months
  Surface EMG
Range of motion of the wrist assess by goniometer and goniometer app | 6 months
  Goniometer and goniometer app

SECONDARY OUTCOMES:
correlation between range of motion of the wrist assessed by goniometer and goniometer app | 1 day
  To assess the correlation of the range of motion evaluated by universal goniometer and goniometer app

CONTACTS AND LOCATIONS:
Overall Officials: Juan-Carlos Zuil-Escobar, PhD, Principal Investigator — CEU San Pablo University
Locations (1):
- CEU-San Pablo Universtiy, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No